CLINICAL TRIAL: NCT05864014
Title: Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Hetrombopag for the Treatment of Chemotherapy-induced Thrombocytopenia in Adults With Solid Tumors.
Brief Title: Hetrombopag for the Treatment of Chemotherapy-Induced Thrombocytopenia in Adults With Solid Tumors.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8735-301
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chemotherapy-Induced Thrombocytopenia
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hetrombopag (Experimental)
  Interventions: Drug: Hetrombopag
- Hetrombopag plus Placebo (Experimental)
  Interventions: Drug: Hetrombopag plus Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hetrombopag — Hetrombopag
  Arms: Hetrombopag
Drug: Hetrombopag plus Placebo — Hetrombopag plus Placebo
  Arms: Hetrombopag plus Placebo
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of current study is to evaluate the efficacy and safety of hetrombopag for the treatment of chemotherapy-induced thrombocytopenia in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18-75 years of age;
2. Participant with a histologically or cytologically confirmed solid tumor receiving treatment with chemotherapeutic agents;
3. Participant experienced thrombocytopenia and chemotherapy delay;
4. ECOG performance status 0-1;
5. Adequate Liver function; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x ULN for participants without liver metastases or 5.0 x ULN for participant with liver metastases);
6. Adequate renal function; serum creatinine < 1.5 x ULN or eGFR≤60 ml/min（Cockcroft-Gault）

Exclusion Criteria:

1. Participant has any history of hematologic diseases other than chemotherapy-induced thrombocytopenia;
2. Participant has serious bleeding symptoms;
3. History of allergy to the study drug;
4. Participant with HIV;
5. Pregnant or lactating women;
6. Participant has received any experimental therapy within 4 weeks prior to screening
7. Other conditions that may affect participant's safety or trial evaluations per investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of treatment responders. | Randomization up to 80 days

SECONDARY OUTCOMES:
Duration from the commencement of treatment to a platelet count ≥100×109/L; | Randomization up to 30 days
Proportion of subjects who could complete chemotherapy without dose modification and rescue therapy and; | Randomization up to 160 days
Proportion of subjects without serious bleeding events; | Randomization up to 190 days
Number of adverse events (AEs)/serious adverse events (SAEs) | Randomization up to 190 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Tumor Research Center of Harbin First Hospital, Haerbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided